CLINICAL TRIAL: NCT07398053
Title: General Practitioner & Pharmacist Support for Discontinuing Long-term Antidepressants in Clinically Stable Patients: a Cluster Randomised Pragmatic Trial in Primary Care
Brief Title: General Practitioner & Pharmacist Support for Discontinuing Long-term Antidepressants in Clinically Stable Patients
Acronym: GPS-AD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University of Liege (Other); Université Catholique de Louvain (Other); Université Libre de Bruxelles (Other); KU Leuven (Other); Universiteit Antwerpen (Other); VUB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2025-0571; KCE-24 1543 (Other Grant/Funding Number: KCE Trials)
Record Dates: First submitted 2025-12-24; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Deprescribing; Antidepressant; Depression Disorder; Discontinuation; Primary Care
Keywords: deprescribing; discontinuation; tapering; depression; antidepressants; long-term use; chronic use; medication review; primary care
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Pragmatic cluster-randomized trial in Belgian primary care. General practitioner (GP) practices are the unit of randomization (cluster) to minimize contamination; patients are the unit of analysis.
Masking Description: Due to the nature of the intervention, participants/clinicians are not blinded. Outcome assessors and statisticians will remain blinded to group allocation until all analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPS-AD intervention (Experimental): The GPS-AD intervention is a structured collaboration between GPs and community pharmacists designed to support the safe discontinuation of long-term AD use in clinically stable adults. The intervention incorporates behavioural activation, motivational support, shared decision-making, personalised tapering schedules, and collaborative care. It follows a stepped-care model and clearly defines the roles of both the GP and pharmacist.
  Interventions: Behavioral: GPS-AD intervention
- care as usual (No Intervention): The management and follow-up in the usual care arm is at the discretion of GP/pharmacist/patient, following the Belgian depression guideline. Patients in the control group will receive care as usual.

INTERVENTIONS:
Behavioral: GPS-AD intervention — The GPS-AD intervention is a structured collaboration between GPs and community pharmacists designed to support the safe discontinuation of long-term AD use in clinically stable adults. The intervention incorporates behavioural activation, motivational support, shared decision-making, personalised tapering schedules, and collaborative care. It follows a stepped-care model and clearly defines the roles of both the GP and pharmacist.
  It starts with an invitation letter and educational brochure that encourages patients to book an appointment with their GP to review their AD use. This is followed by at least one consultation with the GP to discuss the option of tapering AD. If the patient is ready, a personalised tapering plan will be started in collaboration with the pharmacist. The pharmacist provides an initiation consultation, including medication review, tapering plan, potential withdrawal symptoms, motivational support, and a closing consultation focused on future coping.
  Other Names: AD discontinuation; AD deprescribing
  Arms: GPS-AD intervention

SUMMARY:
In Belgium, many adults who have suffered from depression keep using antidepressants on a daily basis for years afterwards, sometimes longer than guidelines recommend. Yet for some people who have been feeling well for a long time, this is no longer necessary, while the continued use of antidepressants can lead to side effects and causes additional costs for the healthcare system.

However, reducing the doses of antidepressants or stopping altogether is not always easy. Some patients are afraid that their depression will return, and GPs and pharmacists often find the subject difficult to broach.

This is why the GPS-AD study is investigating a new approach in which GPs and pharmacists work more closely together to provide better support to patients. First, the GP invites patients who have been taking antidepressants for a long time for a consultation. Together, they discuss whether tapering of the medication is reasonable and feasible. If they agree to stop the treatment, the GP draws up a tapering plan tailored to the patient. The pharmacist helps monitor this process, offering advice and support to the patient while the doses are gradually reduced.

The study will extend over a period of two years and will take place in GP practices throughout Belgium. The new approach based on closer collaboration between GPs and pharmacists will be compared to the current standard of care, to determine whether it helps more long-term users to stop taking antidepressants without experiencing a recurrence of depressive symptoms.

The name of the study, GPS-AD (General Practitioner and Pharmacist Support for Antidepressant Discontinuation), refers to the collaboration between GPs and pharmacists in tapering of antidepressants, and also symbolises the support and guidance (the 'GPS') provided to patients and healthcare providers in assessing whether long-term use of antidepressants is still necessary.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion in the study if they meet all of the following criteria:

* Are 18 years or older and capable of providing informed consent.
* Have their Global Medical File (GMD) managed by one of the participating GPs.
* Have been prescribed AD (any type) by their GP for the treatment of depression, with:

  * at least 6 months of continuous daily use following a first depressive episode, or
  * at least 2 years of continuous daily use in the context of a relapsed depression/recurrent episode
* Are judged by their GP as no longer meeting the criteria for a current depressive disorder.

Exclusion Criteria:

Patients will be excluded from participation in the study if they meet any of the following criteria:

* AD discontinuation is considered contra-indicated by the treating GP.
* The patient is judged by the GP to be at high risk of relapse. This includes any of the following:

  * Current significant depressive symptoms, defined as a score of ≥12 on the PHQ-9
  * Current significant anxiety symptoms, defined as a score of ≥10 on the Generalised Anxiety Disorder-7 (GAD-7) scale.
  * Current suicidal ideation, defined as a score >0 on item 9 (suicidality) of the PHQ-9.
  * The patient is currently receiving only psychiatric treatment (out- or inpatient) for depression

In addition to the criteria increasing the risk of relapse, the following will also be an exclusion criteria:

* The patient has a current psychiatric comorbidity (e.g. bipolar disorder, psychosis, substance use)
* The patient has a diagnosis of dementia or significant cognitive impairment (assessed by GP judgement) or is living in a nursing home.
* The AD is prescribed for a primary indication other than depression, such as anxiety alone without comorbid depressive disorder, or chronic pain.
* The patient has insufficient language proficiency in Dutch or French to participate in the study procedures (e.g. providing consent, completion of questionnaires, interviews).
* use of trazodon as AD as this is mainly used for sleep problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
AD discontinuation (superiority) | 12 months post-randomisation
  Proportion of participants who have stopped antidepressant medication for ≥2 consecutive months at the 12-month follow-up assessment, based on participant self-report.
  This is a binary measure (yes/no).
Depressive symptom severity (inferiority) | 12 months post-randomisation
  PHQ-9 total score (range 0-27; higher scores indicate more severe depressive symptoms) at 12 months post-randomisation; this is a continuous metric. Difference in baseline-corrected mean between groups will be evaluated, with 95% CI. Non-inferiority will be assessed using a prespecified non-inferiority margin of 2 points.
  In this trial, we use co-primary endpoints. The trial will conclude effectiveness only if (1) discontinuation is superior and (2) PHQ-9 is non-inferior.

SECONDARY OUTCOMES:
AD discontinuation | 6, 18 and 24 months post-randomisation
  Proportion of participants who have stopped antidepressant medication for ≥2 consecutive months at the 6-month follow-up assessment, based on participant self-report.
  This is a binary measure (yes/no) at 6, i.e. short-term, 18 and 24, i.e. long-term, months.
Depressive symptom severity | 6, 18 and 24 months post-randomisation
  PHQ-9 total score
Suicidal ideation | 6, 12, 18, and 24 months
  Patient-reported suicidal ideation assessed using item 9 of the Patient Health Questionnaire-9 (PHQ-9), scored 0-3, with higher scores indicating more frequent suicidal thoughts.
Health-related quality of life | 6, 12, 18 and 24 months
  Health-related quality of life measured using the EQ-5D-5L questionnaire, summarized as a country-specific index value derived from the five dimensions
Mental wellbeing | 6, 12, 18, and 24 months post-randomisation
  Mental wellbeing assessed using the Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS), with higher total scores indicating better mental wellbeing.

OTHER OUTCOMES:
Safety: adverse effects of AD | 6, 12, 18, 24 months post-randomisation
  Patient-reported adverse effects of antidepressants assessed using the Antidepressant Side-Effect Checklist (ASEC). The ASEC includes 21 predefined side effects
Safety: relapse or new depressive episode | 6, 12, 18 and 24 months post-randomisation
  Occurrence of relapse or new depressive episode during the preceding 6 months, assessed by the GP based on clinical evaluation and electronic health record review (Yes/No).
Safety: withdrawal symptoms | 6 and 12 months
  Patient-reported antidepressant withdrawal symptoms assessed using an abbreviated version of the Discontinuation Emergent Signs and Symptoms (DESS) questionnaire.
Safety: clinician-assessed withdrawal symptoms | 6 and 12 months post-randomisation
  GP-reported occurrence of antidepressant withdrawal symptoms during the preceding 6 months, based on clinical evaluation and electronic health record review (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Van Leeuwen, MD, PhD, Principal Investigator — University Ghent

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Trial page created by funder: KCE Trials — https://kce.fgov.be/en/kce-trials/funded-trials/gps-ad-general-practitioner-pharmacist-support-for-discontinuing-long-term-antidepressants-in